CLINICAL TRIAL: NCT02679313
Title: Effect of Lens Presentation on the Clinical Oculomotor Assessment at Near
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant is most accurate for this study.
Sponsor: State University of New York College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: Phoropter Study
Record Dates: First submitted 2016-02-01; First posted 2016-02-10 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phoropter (Experimental): Each subject will be tested on 3 separate occasions using either the manual phoropter (American Optical 11625), electronic phoropter (Topcon CV-5000) or the wearable adaptive refractor (VisionFit).
  Interventions: Device: Phoropter

INTERVENTIONS:
Device: Phoropter — Each subject will be tested on 3 separate occasions using either the manual phoropter (American Optical 11625), electronic phoropter (Topcon CV-5000) or the wearable adaptive refractor (VisionFit). Oculomotor measurements, i.e., heterophoria, vergence ranges, AC/A and accommodative findings will be measured at each session using the different devices. Each session will be separated by a minimum of 24 hours and a maximum of 14 days.

SUMMARY:
This study will compare near clinical oculomotor parameters (heterophoria, vergence ranges, AC/A and accommodative findings) measured when lenses and/or prisms are introduced using three different instruments namely: (i) a standard manual phoropter, (ii) an electronic phoropter and (iii) a wearable adaptive refractor (VisionFit).

DETAILED DESCRIPTION:
Previous studies have demonstrated differences in a number of near oculomotor parameters [e.g., heterophoria, accommodative convergence to accommodation (AC/A) ratio] when measured in a manual phoropter versus a trial frame. These differences may be due to variations in proximal vergence, differences in head and eye position and restriction of the peripheral visual field. Further, a number of standard clinical oculomotor procedures require the use of Risley rotary prisms. While prism is typically introduced in a smooth, ramp-like fashion with manual phoropters, step changes in prism are created with electronic phoropters. The precise effect of these variations on clinical measurements is unclear. Accordingly, after a routine refractive examination, a standard clinical near assessment (comprising near heterophoria, AC/A ratio, horizontal vergence ranges, amplitude of accommodation and negative and positive relative accommodation) will be carried out on the same individuals through: (i) a standard manual phoropter (American Optical model 11625), (ii) an electronic phoropter (Topcon CV-5000) and (iii) a wearable adaptive refractor (VisionFit). The latter resembles a trial frame mounted on a helmet carrier (similar to a binocular indirect ophthalmoscope headset) but includes adaptive lenses that can be changed electronically.

ELIGIBILITY:
Inclusion Criteria:

* Corrected visual acuity of at least 20/20 (logMAR = 0.0) or better in each eye

Exclusion Criteria:

* Strabismus, amblyopia, manifest ocular disease.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Near horizontal heterophoria | approximately 15 minutes
  Near horizontal heterophoria (measured in prism diopters) will be recorded using both the Von Graefe and Modified Thorington techniques using each of the three lens presentation devices. The single set of measurements will be recorded approximately 15 minutes after the start of the trial.
Accommodative convergence to accommodation (AC/A) ratio | approximately 15 minutes
  The AC/A ratio will be calculated from measurements of near horizontal heterophoria (quantified in prism diopters) will be recorded using the Modified Thorington technique at 3 different accommodative stimulus levels (1.5D, 2.5D and 3.5D). Measurements will be obtained using each of the three lens presentation devices and calculated in units of prism diopter per diopter accommodation.The single set of measurements will be recorded approximately 15 minutes after the start of the trial.
Horizontal near vergence ranges | approximately 15 minutes
  Near base-in and base-out vergence ranges will be measured (in prism diopters) while the subject fixates a near target. Measurements will be expressed in terms of the blur point, break point and recovery measurement .The single set of measurements will be recorded approximately 15 minutes after the start of the trial.
Minus lens amplitude of accommodation | approximately 15 minutes
  Minus lens amplitude of accommodation (measured in diopters) will be recorded using each of the three lens presentation devices.The single set of measurements will be recorded approximately 15 minutes after the start of the trial.

SECONDARY OUTCOMES:
Negative and Positive Relative Accommodation (NRA and PRA) | approximately 15 minutes
  NRA and PRA (measured in diopters) will be recorded using each of the three lens presentation devices.The single set of measurements will be recorded approximately 15 minutes after the start of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rosenfield, MCOptom, PhD, Principal Investigator — State University of New York College of Optometry
Locations (1):
- SUNY College of Optometry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No